CLINICAL TRIAL: NCT04942054
Title: A Phase 1 Study to Determine Safety, Tolerability, Pharmacokinetics, Pharmacodynamics and Preliminary Efficacy of SCO-120 in Hormone Receptor Positive, HER-2 Negative Advanced Breast Cancer Patients
Brief Title: A Study in Patients With Advanced Breast Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The decision to close is due commercial reasons only
Sponsor: Sun Pharma Advanced Research Company Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SCO-120-19-22
Record Dates: First submitted 2021-06-11; First posted 2021-06-28 (Actual); Last update posted 2023-05-22 (Actual); Status verified 2023-05

CONDITIONS: HER2-negative Breast Cancer; Advanced Breast Cancer; Hormone Receptor-positive Breast Cancer

STUDY DESIGN:
Intervention Model Description: This is a 3 X 3 Design, sequential doses of 300 mg, 600 mg, 800 mg, 1200 mg will be studied. Other dose strength will be studied based on results.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- SCO-120 (Experimental)
  Interventions: Drug: Part 1; Drug: Part 2; Drug: Part 3

INTERVENTIONS:
Drug: Part 1 — Dose escalation cohort
Drug: Part 2 — Pharmacodyanamic (PD) dose exploration cohorts
Drug: Part 3 — Dose expansion at dose(s) ≤ maximum tolerated dose (MTD) cohort

SUMMARY:
A Phase 1, Open label, Dose escalation and Dose expansion study of SCO-120 in HR +ve HER2-ve advanced/ metastatic breast cancer (MBC) patients to evalaute the safety, tolerability and prelimnary efficacy. Initial part with dose escalation is to determine the MTD and RP2D, and PK and PD characterisation. RP2D will be further evalauted for prelimnary efficacy in MBC patients with tretament failure on Aromatase Inhibitor/Fulvestrant/CDK4-6 inhibitors with or with out ESR1 mutation.

DETAILED DESCRIPTION:
Part 1 & 2: Approximately 51 subjects will be enrolled Part 3: Approximately 90 subjects will be enrolled

ELIGIBILITY:
Inclusion Criteria:

1. All 3 parts of Study:

   * Male or females, Age 18 years or older
   * Histologically or cytologically diagnosed with ER+/HER2- adenocarcinoma of the breast cancer with an evidence of metastatic/loco-regionally recurrent disease/unresectable advanced disease not amenable to treatment with curative intent
   * Documentation of ER-positive, HER2-negative status determined based on a biopsy performed at or after diagnosis of local or metastatic recurrence, utilizing an assay consistent with local standards
   * Not more than 3 prior chemotherapeutic regimens
   * ECOG performance status 0-1.
   * Resolution of all adverse events of prior therapy or surgical procedures to National Cancer Institute (NCI) CTCAE v 5.0 Grade ≤1 (except alopecia)
   * Adequate organ and immune system function as indicated by laboratory values
   * Patients of childbearing potential must practice an acceptable method of birth control as judged by the Investigator
   * Female subjects must be non-lactating and non-breast feeding
   * Male subjects should not father a child and must practice an acceptable method of birth control measures Willing and available to participate for the entire study
   * Willing and able to comply with protocol requirements
2. For Part 1& 2:

   * Patient must have evaluable disease (according to RECIST 1.1).
   * Documented disease progression or resistance to at least 1 prior endocrine therapy (with or without CDK 4/6 therapy).
3. For Part 3

   * Patient must have measurable lesions (according to RECIST 1.1)
   * Part 3a: HR+ve, HER2- MBC patients with ESR1 mutations, resistance to atleast one priro endocrine therapy
   * Part 3b: HR+ve HER2- MBC patients resistant to atleast one priro endocrine therapy
   * Part 3c: HR+ve HER2- MBC patients resistant to atleast one priro endocrine therapy, disease progression on Fulvestrant and CDK4/6i
   * Part 3d: Brain metastases secondary to ER+ve HER-ve Breast Cancer:

Measurable brain lesion (≥ 1) as per RANO-BM Criteria, Tretament naive/ Treated- Stable/ Not requiring immediate local therapy known/ Suspected leptomeningeal disease on Stable corticosteriod dose for 7 days prior screeing

Exclusion Criteria:

1. All 3 parts of Study

   * Major surgery <4 weeks of C1D1
   * Evidence of organ dysfunction or inadequate bone marrow reserve or any clinically significant finidngs
   * Patients with visceral crisis or impending visceral crisis and rapidly progressing disease
   * Serology tests +ve for HIV, HCV, HBsAg
   * Inability to swallow oral medication
   * H/o any relevant allergy/hypersensitivity/idiosyncrasy to drugs/ chemically related to Study drug or its excipients
   * Received an IMP within 30 days/5 half life to C1D1
   * Prior treatment with other oral SERDs
   * Use of concomitant medication that might reasonably influence the results or interpretation of the study
   * Requires concurrent systemic anticancer treatment at any time during the study treatment period
   * Known or suspected history of significant drug abuse/Alcohol as judged by the Investigator
   * Known or suspected history of excessive intake of alcohol in the 12 months prior to study entry
   * Malabsorption syndrome/IBD/other illness that would affect oral absorption of Study drug
   * Uncontrolled intercurrent illness that would limit compliance with study requirements / have impact on endpoints / safety
   * ≤6 months H/o MI/unstable angina, ongoing > G2 cardiac dysrhythmia, prolonged QTcF/ uncontrolled AF, coronary/peripheral artery bypass graft, HF of NYHA_Class II or greater and CVA (+TIA)
   * H/o Endometrial intraepithelial neoplasia, other malignancy < 5 yrs prior to enrollment
   * Known active uncontrolled or symptomatic Central Nervous System (CNS) metastases, or leptomeningeal disease as indicated by clinical symptoms (not applicable to Part 3d), carcinomatous meningitis, cerebral edema, and/or progressive growth or pulmonary lymphangitic metastases.
   * Current abnormal vaginal bleeding or symptomatic endometrial disorders.
2. For Part 2: Use of other ET that block the estrogen receptor: atleast 8 weeks before enrollment (28 weeks for fulvestrant) For Part 2: Liver-only metastases (are not evaluable by FES-PET/CT imaging)
3. For Part 3: Any brain lesion requiring immediate local therapy (which includes but is not limited to WBRT, SRS, or surgical resection, for treatment of brain metastases) Requires increase in the dose of corticosteroids for control of CNS symptoms due to brain metastases Poorly controlled (> 2 per month ) generalized or complex partial seizures Who are taking concurrent enzyme-inducing antiepileptic drugs (EIAED) Who has evidence of significant (ie, symptomatic) intracranial haemorrhage Contra indications for repeated MRI assessments

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2022-05-20 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-02-28 (Actual)

PRIMARY OUTCOMES:
Incidence of dose limiting toxicities at each dose levels (Part 1 only) | 28 Days/End of Cycle 1
Incidence and severity of adverse events with each dose level | upto 30 days of last dose
  The intensity of adverse events will be graded as per CTCAE, Version 5.0 and categorized as serious adverse events or non-serious adverse events.

SECONDARY OUTCOMES:
evaluation of Cmax (Part 1 and Part 2) | Through Cycle 1 and Cycle 2 (Each cycle of 28 Days)
  Pharmacokinetic analysis will be performed using non-compartmental analysis. The actual elapsed time from dose will be used in the final pharmacokinetic parameter calculations
evaluation of tmax (Part 1 and Part 2) | Through Cycle 1 and Cycle 2 (Each cycle of 28 Days)
  Pharmacokinetic analysis will be performed using non-compartmental analysis. The actual elapsed time from dose will be used in the final pharmacokinetic parameter calculations
evaluation of AUC (Part 1 and Part 2) | Through Cycle 1 and Cycle 2 (Each cycle of 28 Days)
  Pharmacokinetic analysis will be performed using non-compartmental analysis. The actual elapsed time from dose will be used in the final pharmacokinetic parameter calculations
tumour response | Every 8 weeks, for 'Time point Response (Partial Response[PR], Stable Disease[SD], Disease progression [DP] or Complete Response [CR]), Through study completion, an average of 1 year.

OTHER OUTCOMES:
pharmacodynamic biomarker | At Screening and End of Cycle 1' (Each Cycle of 28 days)
  Pharmacodynamic Biomarkers [Estrogen receptor (ER) expression, Ki67 down regulation from Tissue Biopsy, and Estrogen receptor occupancy with [(18)F] Fluoroestradiol Positron Emission Tomography (18F-FES PET) scan]

CONTACTS AND LOCATIONS:
Locations (6):
- United States (2):
  - Hoag Memorial Hospital Presbyterian, Newport Beach, California
  - The University of Chicago, Chicago, Illinois
- India (4):
  - HealthCare Global Enterprises Ltd, Bangalore, Karnataka
  - HCG Manavata cancer Centre, Nashik, Maharashtra
  - LMMF's Deenanath Mangeshkar Hospital & Research Centre, Pune, Maharashtra
  - Noble Hospital Pvt. Ltd.,, Pune, Maharashtra

IPD SHARING:
Plan to Share IPD: No